CLINICAL TRIAL: NCT05979519
Title: Fresh Carts for Mom's to Improve Food Security and Glucose Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alison Gustafson (Other)
Collaborators: Instacart Health (Unknown); Kentucky Association of Health Plans (Unknown)
Responsible Party: Sponsor-Investigator, Alison Gustafson, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 86500
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy; Type 2 Diabetes Mellitus
Keywords: Pregnancy; Food Insecurity; Food As Medicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Food; Dosage Forms; myotubularin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Grocery Prescription Program (Experimental): Those randomized to the Grocery Prescription intervention will receive the Fresh Funds for Mom's through Instacart immediately
  Interventions: Behavioral: Fresh Funds for Mom's
- Standard Medical Care (Active Comparator): the delayed control group will receive their usual care through their healthcare provider and then participate in Fresh Funds or MTM after the initial 12-weeks of intervention.
  Interventions: Behavioral: Standard Medical care
- MTM (medically tailored frozen meals) (Experimental): Those randomized to the MTM intervention will receive medically tailored frozen meals from Door Dash
  Interventions: Behavioral: Medically Tailored Frozen Meals

INTERVENTIONS:
Behavioral: Fresh Funds for Mom's — Participants will enroll in Instacart Fresh Funds program. Once enrolled participants will select foods that are eligible in the Fresh Funds to be delivered to their home each week for 12 weeks.
  Those in standard care will maintain usual care with their healthcare provider. The standard care arm after the initial 12-weeks and post intervention survey will then select foods that are eligible in the Fresh Funds to be delivered to their home each week for 12 weeks.
  Other Names: Grocery Prescription Program; Food As Medicine
  Arms: Grocery Prescription Program
Behavioral: Standard Medical care — Those in standard care will maintain usual care with their healthcare provider. The standard care arm after the initial 12-weeks and post intervention survey will then select foods that are eligible in the Fresh Funds to be delivered to their home each week for 12 weeks or be provided the medically tailored meals for 12 weeks.
  Arms: Standard Medical Care
Behavioral: Medically Tailored Frozen Meals — Participants will enroll in the MTM program. Once enrolled participants will receive 10 frozen meals delivered by Door Dash to their home each week for 12 weeks.
  Other Names: MTM; Food As Medicine
  Arms: MTM (medically tailored frozen meals)

SUMMARY:
This study will look at the benefit of decreasing food insecurity and improving glucose control among women who either report gestational diabetes (GDM) at 20-28-weeks or have type 2 diabetes (T2DM) with a confirmed pregnancy. Participants will receive a grocery prescription with delivery through Instacart at the start of the study or after 12 weeks or frozen medically tailored meals delivered from Door Dash. Researchers will compare the grocery prescription program, MTM (medically tailored meals), relative to standard of care to see if the impact on these food as medicine programs can improve glucose control over 12-weeks as compared to standard of care.

DETAILED DESCRIPTION:
Women who have a diagnosis of gestational diabetes (GDM) or type 2 diabetes (T2DM) and who report food insecurity using the Hunger Vital Signs Screener will be recruited to participate in a comparative study across two urban communities. One arm will receive a grocery prescription program from Instacart Health to be spent on eligible healthy food items based on My Diabetes Plate. The other arm will receive 10 frozen medically tailored meals delivered to their door each week. The meals are based on diabetes guidelines and are culturally appropriate. Meals are created by a local nonprofit food pantry, Dare to Care, in Louisville, Kentucky and delivered via a partnership with Door Dash - Project Dash. Women will be recruited initially from a registered nurse who works at the clinic sites. The study team will then enroll participants after eligibility screening and conduct further onboarding into the food as medicine package based on locations.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of gestational diabetes or type 2 diabetes
* answer affirmative to one of two questions on the Hunger Vital Signs
* viable pregnancy
* lives in a service area of Instacart delivery
* has a phone or computer which allows ordering food for delivery

Exclusion Criteria:

* Does not speak English
* Does not have a phone, tablet, or computer to order groceries for Instacart
* Plans to move within the next 3 months

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-04-28 (Actual)

PRIMARY OUTCOMES:
Percentage Change in fasting blood glucose | baseline and post intervention, approximately 12 weeks
  Fasting blood glucose obtained baseline and post intervention (prior to delivery) by the healthcare provider from the medical chart.

SECONDARY OUTCOMES:
Change in food insecurity | baseline and post intervention, approximately 12 weeks
  The USDA 6 item food insecurity screener will be used. The scale ranges from 0 to 6 with a higher score indicating greater food insecurity.
Change in self efficacy | baseline and post intervention, approximately 12 weeks
  The self efficacy scale for diabetes measures the confidence in managing diabetes. Scores range from 1 to 10 with a higher score indicating greater confidence in managing diabetes.
Change in blood pressure | baseline and post intervention, approximately 12 weeks
  Diastolic and systolic Blood pressure will be obtained baseline and post intervention (prior to delivery) by the healthcare provider from the medical chart.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Gustafson, PhD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - U of L Health, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: No